CLINICAL TRIAL: NCT02148822
Title: Visceral Leishmaniasis and Malnutrition in Amhara Regional State, Ethiopia
Acronym: VL&MNEthio
Status: Completed | Type: Observational
Sponsor: Instituto de Salud Carlos III (Other Government)
Collaborators: UBS Optimus Foundation (Other); Armauer Hansen Research Institute, Ethiopia (Other)
Responsible Party: Principal Investigator, Estefania Custodio, Researcher, Instituto de Salud Carlos III
Other Study IDs: Opt1228
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Visceral Leishmaniasis; Malnutrition
Keywords: Visceral leishmaniasis; kala azar; malnutrition; stunting; thinness; Leishmania donovani
MeSH Terms: conditions — Leishmaniasis, Visceral; Malnutrition; Growth Disorders; Thinness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Malnourished: Children with either height for age z score or body mass index for age z score below 2 standard deviations according to the World Health Organization Growth Standards for children younger than 5 years and the 2007 WHO Growth Reference for children of 5 years or older.
- Not malnourished: Children with either height for age z score or body mass index for age z score equal or higher than 2 standard deviations according to the World Health Organization Growth Standards for children younger than 5 years and the 2007 WHO Growth Reference for children of 5 years or older.

SUMMARY:
The project Visceral Leishmaniasis and Malnutrition is a cohort study that aimed to assess the association between malnutrition and visceral leishmaniasis (VL). It was conducted in Libo Kemkem and Fogera districts of the Amhara Regional State in Ethiopia. Clinical, anthropometric, biochemical, immunological, parasitological and sociodemographic data of school age children from VL high prevalence communities were collected in December 2009, May 2010 and February 2011.

ELIGIBILITY:
Inclusion Criteria:

* Reported age between 4 and 15 years of age
* Currently living in the selected household

Exclusion Criteria:

* To be ill of visceral leishmaniasis at the time of the survey
* To be positive to visceral leishmaniasis infection tests at the time of the first survey
* To be under treatment for visceral leishmaniasis at the time of the survey
* To be extremely ill of any other condition

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: School age children from VL high prevalent communities of Libo Kemkem and Fogera districts in Amhara Regional State, Ethiopia
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2009-12; Primary Completion 2009-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
visceral leishmaniasis disease | December 2009, May 2010 and February 2011 (up to 14 months)

SECONDARY OUTCOMES:
visceral leishmaniasis infection | December 2009, May 2010 and February 2011 (up to 14 months)

OTHER OUTCOMES:
Growth | December 2009, May 2010 and February 2011 (up to 14 months)

CONTACTS AND LOCATIONS:
Overall Officials: Estefania D Custodio, PhD, Study Chair — Instituto de Salud Carlos III

REFERENCES:
- [Result] Lopez-Perea N, Sordo L, Gadisa E, Cruz I, Hailu T, Moreno J, Aseffa A, Canavate C, Custodio E. Knowledge, attitudes and practices related to visceral leishmaniasis in rural communities of Amhara State: a longitudinal study in northwest Ethiopia. PLoS Negl Trop Dis. 2014 Apr 17;8(4):e2799. doi: 10.1371/journal.pntd.0002799. eCollection 2014 Apr. PMID 24743328
- [Result] Custodio E, Gadisa E, Sordo L, Cruz I, Moreno J, Nieto J, Chicharro C, Aseffa A, Abraham Z, Hailu T, Canavate C. Factors associated with Leishmania asymptomatic infection: results from a cross-sectional survey in highland northern Ethiopia. PLoS Negl Trop Dis. 2012;6(9):e1813. doi: 10.1371/journal.pntd.0001813. Epub 2012 Sep 27. PMID 23029576
- [Result] Sordo L, Gadisa E, Custodio E, Cruz I, Simon F, Abraham Z, Moreno J, Aseffa A, Tsegaye H, Nieto J, Chicharro C, Canavate C. Low prevalence of Leishmania infection in post-epidemic areas of Libo Kemkem, Ethiopia. Am J Trop Med Hyg. 2012 Jun;86(6):955-8. doi: 10.4269/ajtmh.2012.11-0436. PMID 22665599
- [Result] Custodio E, Descalzo MA, Roche J, Molina L, Sanchez I, Lwanga M, Torres AM, Fernandez-Zincke E, Bernis C, Villamor E, Baylin A. The economic and nutrition transition in Equatorial Guinea coincided with a double burden of over- and under nutrition. Econ Hum Biol. 2010 Mar;8(1):80-7. doi: 10.1016/j.ehb.2009.10.001. Epub 2009 Oct 31. PMID 19959405
- [Derived] Herrador Z, Perez-Formigo J, Sordo L, Gadisa E, Moreno J, Benito A, Aseffa A, Custodio E. Low Dietary Diversity and Intake of Animal Source Foods among School Aged Children in Libo Kemkem and Fogera Districts, Ethiopia. PLoS One. 2015 Jul 23;10(7):e0133435. doi: 10.1371/journal.pone.0133435. eCollection 2015. PMID 26203904